CLINICAL TRIAL: NCT02905799
Title: Evolution of Pain at Three Months by Oral Resveratrol in Primary Knee Osteoarthritis: a Multicenter, Double-blind, Randomized, Placebo-controlled Trial
Brief Title: Resveratrol in Knee Osteoarthritis
Acronym: ARTHROL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: P150938; 2016-A01310-51 (Registry Identifier: ANSM)
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Knee; Resveratrol; Oral Treatment; Pain; Trial
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral resveratrol (Experimental): Resveratrol will be administered orally, at the dose of 40 mg (2 caplets) twice a day for one week, then at the dose of 20 mg (1 caplet) twice a day, for a total duration of 6 months.
  Interventions: Drug: oral resveratrol
- Oral Placebo (Placebo Comparator): Placebo will be administered orally : 2 caplets twice a day for one week, then 1 caplet twice a day, for a total duration of 6 months.
  Interventions: Drug: oral placebo

INTERVENTIONS:
Drug: oral resveratrol — Resveratrol will be administered orally, at the dose of 40 mg (2 caplets) twice a day for one week, then at the dose of 20 mg (1 caplet) twice a day, for a total duration of 6 months.
  Arms: Oral resveratrol
Drug: oral placebo — Placebo will be administered orally : 2 caplets twice a day for one week, then 1 caplet twice a day, for a total duration of 6 months
  Arms: Oral Placebo

SUMMARY:
The purpose of this study is to determine whether resveratrol is effective in the treatment of painful knee osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the first cause of handicap in individuals over 40 years-old in France. OA physiopathology is driven in part by local joint inflammation responsible for pain and joint destruction. Experimental studies have shown that resveratrol, a molecule antagonist to the aryl hydrocarbon receptor, has anti-inflammatory and chondroprotective properties in vitro and in vivo. The investigators hypothesize that oral resveratrol, in a new formulation improving its bioavailability, could reduce knee pain at 3 months as compared with placebo in people with knee OA.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years-old
* Knee osteoarthritis fulfilling 1986 American College of Rheumatology (ACR) criteria
* Pain on numeric rating scale ≥ 40/100
* Symptom duration ≥ 1 month
* Kellgren and Lawrence X-Ray score 1, 2 or 3
* Written consent obtained
* Health insurance cover

Exclusion Criteria:

* History of symptomatic crystal or inﬂammatory arthritis
* Knee surgery ≤ 1 year
* Knee trauma ≤ 2 months
* Knee intra-articular injections of corticosteroids and/or hyaluronic acid ≤ 2 months
* Neurologic disorders involving the lower limbs
* Patient not understanding and not speaking french
* Participation in another biomedical research
* Contraindication to resveratrol or hypersensitivity to any of its constituents
* Current use of intramuscular, intravenous or oral corticosteroids
* Uncontrolled diseases that may require intramuscular, intravenous or oral corticosteroids
* Current use of anticoagulants

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-05-12 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in knee pain in the previous 48 hours | at 3 months
  Using a self-administered 11-point pain numeric rating scale, with 0 = no pain and 100 = maximal pain

SECONDARY OUTCOMES:
Mean change from baseline in knee pain in the previous 48 hours | at 6 months
  Using a self-administered 11-point pain numeric rating scale, with 0 = no pain and 100 = maximal pain
Mean change from baseline in specific activity limitation | at 3 months
  Using self-administered WOMAC function subscore, with 0 = no
Mean change from baseline in specific activity limitation | at 6 months
  Using self-administered WOMAC function subscore, with 0 = no
Mean change from baseline in patient's global assessment | at 3 months
  Using a self-administered 11-point global assessment numeric rating scale, with 0 = worst possible and 100 = best possible
Mean change from baseline in patient's global assessment | at 6 months
  Using a self-administered 11-point global assessment numeric rating scale, with 0 = worst possible and 100 = best possible
Proportion of OARSI-OMERACT responders | at 3 months
  OARSI-OMERACT response
Proportion of OARSI-OMERACT responders | at 6 months
  OARSI-OMERACT response
Number of intra-articular injections of corticosteroids or hyaluronic acid since last contact | at 3 months
  using self-reporting
Number of intra-articular injections of corticosteroids or hyaluronic acid since last contact | at 6 months
  using self-reporting
Self-reported consumption of analgesics (non-opioid, weak and strong opioids) since last contact | at 3 months
  using a self-administered 4-class scale (never, several times a month, several times a week, daily)
Self-reported consumption of analgesics (non-opioid, weak and strong opioids) since last contact | at 6 months
  using a self-administered 4-class scale (never, several times a month, several times a week, daily)
Self-reported consumption of non-steroidal anti-inflammatory drugs since last contact | at 3 months
  using a self-administered 4-class scale (never, several times a month, several times a week, daily)
Self-reported consumption of non-steroidal anti-inflammatory drugs since last contact | at 6 months
  using a self-administered 4-class scale (never, several times a month, several times a week, daily)

CONTACTS AND LOCATIONS:
Overall Officials: Christelle NGUYEN, MD, PhD, Study Director — Université Paris Descartes, PRES Sorbonne Paris Cité
Locations (3):
- France (3):
  - Rheumatology Department, Saint Antoine Hospital, Paris, paris
  - Rehabilitation Department, Cochin Hospital, Paris, Paris
  - Rehabilitation department , CHU Clermont-Ferrand, Cébazat

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nguyen C, Coudeyre E, Boutron I, Baron G, Daste C, Lefevre-Colau MM, Sellam J, Zauderer J, Berenbaum F, Rannou F. Oral resveratrol in adults with knee osteoarthritis: A randomized placebo-controlled trial (ARTHROL). PLoS Med. 2024 Aug 13;21(8):e1004440. doi: 10.1371/journal.pmed.1004440. eCollection 2024 Aug. PMID 39137167
- [Background] Nguyen C, Boutron I, Baron G, Coudeyre E, Berenbaum F, Poiraudeau S, Rannou F. Evolution of pain at 3 months by oral resveratrol in knee osteoarthritis (ARTHROL): protocol for a multicentre randomised double-blind placebo-controlled trial. BMJ Open. 2017 Sep 29;7(9):e017652. doi: 10.1136/bmjopen-2017-017652. PMID 28965100